CLINICAL TRIAL: NCT04024358
Title: A New Scoring System for Perineural and Vascular Invasion in Pancreatic Cancer
Acronym: VANISSh
Status: Active, not recruiting | Type: Observational
Sponsor: Massimo Falconi (Other)
Responsible Party: Sponsor-Investigator, Massimo Falconi, Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: VANISSh
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Pancreas Cancer
Keywords: neural invasion; vascular invasion
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

SUMMARY:
The aim of this study is to validate both retrospectively and prospectively a newly proposed scoring system for perineural and vascular invasion in pancreatic ductal cancer and correlate it with disease free survival, early recurrence, site of recurrence, overall survival and neoadjuvant treatment.

DETAILED DESCRIPTION:
Perineural invasion (PNI) is defined as the presence of cancer cells along nerves and/or within the epineural, perineural and endoneural spaces of the neuronal sheath.Clinically, PNI is associated with increased tumor recurrence, poor survival after pancreatectomy and pain, an invalidating symptom that may impair quality of life. Pancreatic ductal adenocarcinoma has one of the highest incidences of PNI (70-100%) among all types of cancer, which correlates with a poor prognosis and decreased survival. PNI is a still not uniformly characterized or quantified event, usually it is described only dichotomously ("present" or "absent"), despite some efforts to use a more detailed scoring system. However, these scores are not specifically developed for pancreatic surgical specimen. Vascular invasion (VI), which is assumed to be associated with a more aggressive tumor biology and dissemination, lacks a specific scoring system as well. The primary aim of this study is to validate both retrospectively and prospectively a novel PNI and VI scoring system aimed at a more detailed stratification of perineural invasion, together with an accompanying scoring system for vascular invasion, and correlated them with disease free survival (DFS).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients undergoing all types of pancreatic resection (pancreatoduodenectomy, left pancreatectomy, total pancreatectomy, both laparotomic and laparoscopic).
* Proven pancreatic ductal adenocarcinoma (cytology or biopsy).
* Patients that received neoadjuvant therapy (CT +/- RT) can be included.
* Patients able to sign the informed consent.

Exclusion Criteria:

* Age < 18 years.
* Patients with other ongoing oncological diseases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed pancreatic ductal adenocarcinoma at the histological examination after surgery with resective purposes.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
PNI and VI correlation with DFS | Up to 36 months
  Analyze if the severity of perineural and perivascular invasion correlates with disease free survival

SECONDARY OUTCOMES:
PNI and VI correlation with other clinical variables | Up to 6 years
  Analyze if the severity of perineural and perivascular invasion correlates with major clinical variables such as early recurrence, site of recurrence, overall survival.
PNI and VI correlation with neoadjuvant treatment | Up to 12 months
  Analyze if neoadjuvant treatment impacts the severity of perineural and perivascular invasion.
Correlation of neurotoxicity with PNI | Up to 12 months
  For patients undergoing chemotherapeutic treatment, correlate (if experienced) neurotoxic side effects with PNI presence and scoring system to treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Marco Schiavo Lena, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided